CLINICAL TRIAL: NCT01891877
Title: Is Sickle Cell Trait as Benign as is Usually Assumed?
Brief Title: Sickle Cell Trait in Football Players
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of South Florida (Other)
Responsible Party: Principal Investigator, Carroll Flansburg, Research Coordinator, University of South Florida
Other Study IDs: SCT in Football; NCAA (Other: National Collegiate Athletic Association)
Record Dates: First submitted 2013-06-25; First posted 2013-07-03 (Estimated); Last update posted 2014-10-20 (Estimated); Status verified 2014-10

CONDITIONS: Sickle Cell Trait
Keywords: Sickle Cell Trait; Football; Sickling; Heat Illness; SCT
MeSH Terms: conditions — Sickle Cell Trait; Heat Stress Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Buccal swabs will be collected from each participant.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Current or Former Football Players: Any former or current high school or college football players who carries sickle cell trait.

SUMMARY:
This study will look at the five different types of sickle cell and their relation to self-reported ill health to determine whether or not one or two of the sickle cell haplotypes are correlated with worse health outcomes. Participants can do complete the study in under half an hour in the privacy of their own home.

DETAILED DESCRIPTION:
Sickle cell anemia is a disease which results from the inheritance of two hemoglobin S (Hb S) genes. Sickle-cell anemia individuals are referred to as Hb SS patients, and are known to suffer from a variety of life-threatening symptoms. Paramount in the clinical complications of sickle cell patients is the "sickle-cell crisis". If a crisis is not stopped by prompt medical attention, it may result in death. It is becoming increasingly clear that some sickle cell anemic patients have more benign clinical profiles than do others. The genetic reason for such clinical differences has been well determined: although the mutation that changes the "normal" hemoglobin gene is the same in all patients, the genetic material outside of the gene influences how the gene is expressed. This genetic material is referred to as the beta-globin haplotype. Carriers of the sickle cell gene are referred to as Hb AS individuals. Hb AS carriers usually have a normal life free of the clinical problems associated with the disease suffered by sickle cell patients. However, it is becoming increasingly clear that under strenuous situations, some Hb AS carriers do experience heat illness and other life threatening problems while others do not. The purpose of this project is to determine if there is a genetic reason for why some athlete carriers of the sickle cell trait experience heat illness, while others do not. Although the genetic reason for the different clinical outcomes of sickle cell anemic patients is now well understood (different haplotypes result in different disease courses), the possibility that the same haplotypes might be the reason why some sickle cell carriers have worse clinical profiles has never been explored. In this project we will work with a sickle-cell trait registry of athletes, and we will test the haplotypes of Hb AS athletes who have and who have not had heat illness. Our study is the first to attempt to clarify if there is a genetic reason for this occurrence. Total participation time for the study is thirty minutes or less. Information provided by the participant will be analyzed within one year of participation. Deidentified results will be kept for five years, per the University of South Florida's Institutional Review Board protocol, and will be available upon request to the principal investigator. Participants can do complete the study in under half an hour in the privacy of their own home.

ELIGIBILITY:
Inclusion Criteria:

* over the age of 18
* male
* has previously played or currently plays high school or college football
* carries sickle cell trait

Exclusion Criteria:

* under the age of 18
* female
* does not carry sickle cell trait
* has not played or does not play high school or college football

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult males who currently or formerly played high school or college football and know that they carry sickle cell trait.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2012-10; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Poor health outcomes | 30 minutes or less to complete survey and buccal swab
  Any ill health events, such as excessive dehydration, muscle cramping, fatigue, shortness of breath, sickling crises, that can be linked to a sickling event.

CONTACTS AND LOCATIONS:
Overall Officials: Carroll N Flansburg, in progress, Principal Investigator — University of South Florida
Locations (1):
- University of South Florida, Tampa, Florida, United States